CLINICAL TRIAL: NCT02880761
Title: Cohort Study on A Following-up System of Native Arteriovenous Fistulae in Chinese Patients Treated by Maintenance Hemodialysis
Brief Title: Cohort Study on A Following-up System of Native Arteriovenous Fistulae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Peking University International Hospital (Other)
Responsible Party: Principal Investigator, Dongliang Zhang, MD, Associated director of blood purification center, Peking University International Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-019
Record Dates: First submitted 2016-08-17; First posted 2016-08-26 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Arteriovenous Fistulae
Keywords: hemodialysis; chronic renal failure; arteriovenous fistulae
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Punctures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients with AVF will be followed up by a preset following-up system. Interventions would be administered according to the assessment for AVF, which including the surgery and puncture of AVF. For AVF surgery, a certain vein would be used in the operation according to the assessment results. For AVF puncture, the methods, such as 'button hole', 'rope ladder', dwelling needle, would be selected prospectively according to the assessment results.
  Interventions: Procedure: Assessment guiding surgery and puncture for AVF
- Control (No Intervention): Patients in other hemodialysis centers who are treated by routine protocal would be enrolled into control group. Their clinical data would be collected and compared with intervention group.

INTERVENTIONS:
Procedure: Assessment guiding surgery and puncture for AVF — Assessment guiding surgery and puncture for AVF. Assessing the parameters of vascular vessels during following-up and making suggestions on surgery and puncture of AVF
  Arms: Intervention

SUMMARY:
A cohort including more than 100 maintenance hemodialysis patients will be followed up according to a certain Following-up System of Native Arteriovenous Fistulae (AVF) prospectively. The assessment results of the Following-up System of AVF help the physicians make decisions of AVF surgery and puncture methods. The results of this study would identify the effect of the system on survival of AVF. Other 100 hemodialysis patients from other centers will be treated by routine protocol and compared to the experiment goup.

DETAILED DESCRIPTION:
The Following-up System of AVF includes 3 stages. In the 1st stage, before AVF surgery operation, the contents of Following-up System of AVF include history, physical exam, ultrasonography detection. The assesment results will guide the methods of the AVF surgery operation. In the 2nd stage, before AVF puncture firstly and 3 months after AVF operation, the contents of Following-up System of AVF include physical exam and ultrasonography detection. The results will help the nurses and doctors make a decision of the method of AVF puncture. In the 3rd stage, during the following 2 years after AVF puncture successfully, the contents include physical exam and ultrasonography detection regularly. The adequacy of hemodialysis by using AVF will be assessed by urea clearance index (Kt/V).

The data of patients in other hemodialysis centers will be recorded and compared to the patients in experiment group.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance hemodialysis patients using AVF;
* Ages 18-70 years old;
* Agreement with frequent following-up.

Exclusion Criteria:

* Younger than 18 years or elder than 70 years;
* Cachexia;
* Acute renal failure;
* Exceptive life time less than 6 months;
* Pregnant or planning pregnant;
* Waiting for renal transplantation or transferring to peritoneal dialysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2016-07; Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dongliang Zhang, Doctor, Study Chair — Peking University Hospital
Locations (1):
- Peking University International Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Patients with native arterovenous fistula (AVF) will be followed up by a preset following-up system. Interventions would be administered according to the assessment for AVF, which including the surgery and puncture of AVF. For AVF surgery, a certain vein would be used in the operation according to the assessment results. For AVF puncture, the methods, such as 'button hole', 'rope ladder', dwelling needle, would be selected prospectively according to the assessment results.
  Assessment guiding surgery and puncture for AVF: Assessment guiding surgery and puncture for AVF. Assessing the parameters of vascular vessels during following-up and making suggestions on surgery and puncture of AVF
Period: Overall Study
Arm/Group | Intervention | Control
Started | 103 | 106
Completed | 87 | 85
Not Completed | 16 | 21
Not completed — Death | 6 | 8
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Protocol Violation | 4 | 3
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 87 | 85 | 172
Age, Continuous [Mean (Standard Deviation); unit: year] | 55.3 (11.9) | 55.3 (12.1) | 55.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 48 | 98
  Male | 37 | 37 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han | 87 | 85 | 172
Height(cm) [Mean (Standard Deviation); unit: cm] | 167.3 (7.7) | 167.4 (7.9) | 167.3 (7.8)
Weight(Kg) [Mean (Standard Deviation); unit: Kg] | 67.0 (12.5) | 66.6 (10.7) | 66.8 (11.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fistula Failure
Description: The AVF can not be used for hemodialysis treatment 3 months after surgery, which it is defined as Primary Failure of AVF. The primary failure of AVF is regarded as the primary outcome of the patients who were followed up. The ratio of primary failure will be compared between two groups.
Time Frame: 3 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 87 | 85
Participants | 11 | 15

2. Secondary Outcome: Life Time of AVF
Description: The life time of an available AVF since the AVF is functionable. The life time of an AVF is a period time from the AVF used for hemodialysis treatment at first time to the last time when the AVF can not be used for hemodialysis therapy,, whichever came first, assessed up to 48 months. Since the AVF will be punctured in every hemodialysis session, the function of AVF were detected during every treatment session (3 times per week).
Time Frame: Equal to or larger than 2 years
Measure: Mean (Standard Deviation); unit: month
Arm/Group | Intervention | Control
Number analyzed (Participants) | 87 | 85
month | 30.5 (21.6) | 26.8 (19.9)

3. Other Pre Specified Outcome: Mean Value of Urea Clearance Index During 24 Months
Description: As a parameter of hemodialysis adequacy, urea clearance index (Kt/V) will be detected very month. The Kt/V should be larger than 1.2 , which were regarded as being adequate in the hemodialysis session. This parameter will be tested every month and the mean value were be calculated according to the records during 24 months. Those who with Kt/V less than 1.2 for 3 times would be defined as the patient with unfunctional AVF. The values of Kt/V in unfunctional AVF patients would not be used in statistic analysis.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: Kt/V
Arm/Group | Intervention | Control
Number analyzed (Participants) | 87 | 85
Kt/V | 1.31 (.28) | 1.29 (.27)

ADVERSE EVENTS:
Time Frame: 2 years.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 6/103 | 8/106
Serious Adverse Events (participants affected / at risk) | 4/103 | 6/106
Other Adverse Events (participants affected / at risk) | 2/103 | 1/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=103) | Control (N=106)
acute myocardial infarction (Cardiac disorders) | 2 (2) | 5 (5) — Newly happened acute myocardial infarction.
Heart Failure (Cardiac disorders) | 2 (2) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=103) | Control (N=106)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT02880761/Prot_SAP_000.pdf